CLINICAL TRIAL: NCT03157141
Title: Ankle Osteoarthritis and Its Treatments : Impact on Foot & Ankle Biomechanics
Brief Title: Ankle Osteoarthritis
Acronym: AO-IFAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0223
Record Dates: First submitted 2017-03-27; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Ankle Osteoarthritis
Keywords: Ankle osteoarthritis; total ankle replacement; ankle arthrodesis; kinematics; kinetics; plantar pressure measurements; functional compensatory adaptations
MeSH Terms: interventions — Arthroplasty, Replacement, Ankle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group, CG: For the purpose of the study, forty subjects for each group will be recruited. The control group (CG group) (so-called healthy subjects) CG will be recruited following the recruitment of the AA group and of the TAR group, as a sex, age and BMI matched design will be pursued. Inclusion criteria for the CG group are no history of orthopaedic lower limb surgery and absence of any known neurological or systematic disease.
- Total ankle replacement group (TAR group): The number of AA and TAR subjects used in a majority of studies to analyze the functional repercussion of an ankle arthrodesis or a total ankle replacement varied between 10 and 35 subjects.
  Interventions: Procedure: Total ankle replacement
- Ankle arthrodesis group (AA group): The number of AA and TAR subjects used in a majority of studies to analyze the functional repercussion of an ankle arthrodesis or a total ankle replacement varied between 10 and 35 subjects
  Interventions: Procedure: Ankle arthrodesis

INTERVENTIONS:
Procedure: Ankle arthrodesis — Ankle arthrodesis consists of fusioning the joint surfaces of the ankle. The procedure will consist of removing the diseased cartilage and subchondral bone until bleeding of the cancellous bone surfaces is revealed. The bone ends will be opposed in the most appropriate and stable position and stabilized with screws or plates.
  Groups: Ankle arthrodesis group (AA group)
Procedure: Total ankle replacement — A two-component ankle prosthesis will be inserted using the surgeon's standard technique, which essentially involves an anterior approach to the ankle joint. Once the joint is exposed, talar and tibial surfaces will be prepared and the prosthesis will be implanted according to the prosthesis surgical technique and its instrumentation.
  Groups: Total ankle replacement group (TAR group)

SUMMARY:
Ankle osteoarthritis is a progressive degenerative joint disease that is characterized by severe pain, loss of autonomy, diminished health-related quality of life, functional disability and diminished physical ability to fulfill occupational duties of life in its end-stage. Current surgical treatments for ankle osteoarthritis are ankle arthrodesis and total ankle replacement. Despite the good pain relief provided by these procedures, patients are still experiencing post-operatively important functional limitations in their activities of the daily living which affect their independency and quality of life. In order to remain capable of performing primary activities of the daily living, those patients have to make functional compensatory adaptations in the ipsilateral adjacent joints that will cause additional degenerative joint disease in those joints.

Currently, the outcome of foot and ankle surgery is primarily based on clinical, radiographic and questionnaire outcomes. However, these outcome measures have been criticized for not being sensitive enough to detect clinically meaningful change in foot function. To tackle these shortcomings, an advanced clinical examination platform integrating pressure-force-kinematic measurement devices was developed and showed its clinical value for the detection of intrinsic foot mobility impairments. Surprisingly, up-to-now, no study has included this integrated use of three-dimensional multi-segment foot models, plantar pressure platform and a force platform to report on the functional outcome of an ankle arthrodesis or a total ankle replacement.

Therefore, a multi-centre study will be conducted with two foot & ankle surgery centres. Both centres are equipped with the same advanced clinical examination platform. It is believed that proposed approach has the potential to provide further insight in the true functional changes related to ankle arthrodesis and total ankle replacement. This may in turn result in improved rehabilitation, less risk for post-operative complications, earlier discharge and quicker resumption of normal activities of the daily living, which would make ankle arthrodesis and total ankle replacement more cost-efficient and could potentially affect thousands of patients each year. Therefore, the hypotheses of the present study are:

* Hypothesis (H1): Subjects with an ankle arthrodesis require a greater reorganization of foot and lower limb kinematic and kinetic patterns to respond to mechanical requirements of level walking compared to subjects with a total ankle replacement.
* Null hypothesis (H0): Subjects with an ankle arthrodesis do not require a greater reorganization of foot and lower limb kinematic and kinetic patterns to respond to mechanical requirements of level walking compared to subjects with a total ankle replacement.

ELIGIBILITY:
Inclusion Criteria:

* primary osteoarthritis
* post-traumatic osteoarthritis with an aligned or partially reducible deformity of the ankle and/or hindfoot

Exclusion Criteria:

* history of orthopaedic lower limb surgery except for the ankle
* neuromuscular disorders
* vascular insufficiency
* significant skin conditions such as skin ulcers or skin grafts

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from ankle osteoarthritis.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Foot and lower limb kinematics (degrees). | change from baseline (preoperative) to 12 months post-operatively
  The Rizzoli 3D multi-segment foot model and the Rizzoli 3D lower limb model will be used to calculate changes pre-and post-operative foot and lower limb kinematics during barefoot walking.
Foot and lower limb kinematics (degrees). | change from baseline (preoperative) to 24 months post-operatively
  The Rizzoli 3D multi-segment foot model and the Rizzoli 3D lower limb model will be used to calculate changes pre-and post-operative foot and lower limb kinematics during barefoot walking.
Joint moments (N.m/kg) | Change from baseline (preoperative) to 12 months post-operatively
  3D multisegment foot kinetic model will allow to quantify mechanical loading of intrinsic foot joints during barefoot walking.
Joint moments (N.m/kg) | Change from baseline (preoperative) to 24 months post-operatively
  3D multisegment foot kinetic model will allow to quantify mechanical loading of intrinsic foot joints during barefoot walking.
Force-time impulses (N.s) | Change from baseline (preoperative) to 12 months post-operatively
  Force-time impulse is used to evaluate the effectiveness of a treatment at a specific foot location
Force-time impulses (N.s) | Change from baseline (preoperative) to 24 months post-operatively
  Force-time impulse is used to evaluate the effectiveness of a treatment at a specific foot location
Power (W/kg) | Change from baseline (preoperative) to 24 months post-operatively
  3D multisegment foot kinetic model will allow to quantify mechanical loading of intrinsic foot joints during barefoot walking.
Power (W/kg) | Change from baseline (preoperative) to 12 months post-operatively
  3D multisegment foot kinetic model will allow to quantify mechanical loading of intrinsic foot joints during barefoot walking.

SECONDARY OUTCOMES:
Demographic data | pre-operatively
Mechanical axis of the foot and lower limb (degrees) | pre-operatively
  The medical records of participants who are eligible for the study, will be reviewed by a member of the research team to collect the standardized weightbearing anteroposterior ankle Meary view and standardized weightbearing lateral foot (and ankle) view to measure the mechanical axis of the foot and lower limb
Position of the ankle arthrodesis or of the ankle prosthesis (degrees) | Change from baseline (preoperative) to 12 months post-operatively
  The medical records of participants who are eligible for the study, will be reviewed by a member of the research team to collect the standardized weightbearing anteroposterior ankle Méary view and standardized weightbearing lateral foot (and ankle) view to measure the position of the ankle arthrodesis and/or of the ankle prosthesis.
Health-related quality of life (SF-36) | Change from baseline (preoperative) to 12 months post-operatively
  The Short-Form-36 (Version two) (SF-36) questionnaire will be used to assess health-related quality of life. The SF-36 is a 36 question survey that measures eight health concepts most affected by disease and treatment. The eight health concepts can then be used to form two summary measures: physical health and mental health. The SF-36 has been extensively validated and is one of the most widely used instruments to measure health status. The SF-36 has sound reliability and validity
Health-related quality of life (SF-36) | Change from baseline (preoperative) to 24 months post-operatively
  The Short-Form-36 (Version two) (SF-36) questionnaire will be used to assess health-related quality of life. The SF-36 is a 36 question survey that measures eight health concepts most affected by disease and treatment. The eight health concepts can then be used to form two summary measures: physical health and mental health. The SF-36 has been extensively validated and is one of the most widely used instruments to measure health status. The SF-36 has sound reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc BESSE, Dr, Principal Investigator — Centre Hospitalier Lyon-Sud, 69495 Pierre-Bénite Cédex, France
Locations (1):
- Centre Hospitalier Lyon-Sud, Pierre-Bénite, France